CLINICAL TRIAL: NCT01202890
Title: Phase IB Study of Lenalidomide (Revlimid®) With Liposomal Doxorubicin (Doxil®) and Bevacizumab (Avastin®) for Patients With Platinum Resistant Ovarian Cancer.
Brief Title: Study of Revlimid With Doxil and Avastin for Patients With Platinum Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to inadequate rate of accrual.
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1001
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
Keywords: lenalidomide; revlimid; liposomal doxorubicin; doxil; bevacizumab; avastin; platinum resistant ovarian cancer; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Lenalidomide; liposomal doxorubicin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): At the expansion phase: Revlimid 20 mg (days 1-21), Doxil 30 mg/m2 on Day 1 and Avastin 15 mg/kg on Day 1, every 3 weeks. If this regimen is not cumulatively tolerable, Avastin will be administered every other course. Patients will be received up to 6 cycles or disease progression, followed by Revlimid maintenance at 25 mg PO q Day for 3 weeks every 4 weeks in patients with stable disease.
  Interventions: Drug: Lenalidomide, Liposomal Doxorubicin, Bevacizumab; Drug: Revlimid, Doxil, Avastin

INTERVENTIONS:
Drug: Lenalidomide, Liposomal Doxorubicin, Bevacizumab — At the expansion phase: Revlimid 20 mg (days 1-21), Doxil 30 mg/m2 on Day 1 and Avastin 15 mg/kg on Day 1, every 3 weeks. If this regimen is not cumulatively tolerable, Avastin will be administered every other course.
  Patients will be received up to 6 cycles or disease progression, followed by Revlimid maintenance at 25 mg PO q Day for 3 weeks every 4 weeks in patients with stable disease.
  Other Names: Revlimid, Doxil, Avastin
Drug: Revlimid, Doxil, Avastin — At the expansion phase: Revlimid 20 mg (days 1-21), Doxil 30 mg/m2 on Day 1 and Avastin 15 mg/kg on Day 1, every 3 weeks. If this regimen is not cumulatively tolerable, Avastin will be administered every other course. Patients will be received up to 6 cycles or disease progression, followed by Revlimid maintenance at 25 mg PO q Day for 3 weeks every 4 weeks in patients with stable disease.

SUMMARY:
This study will test the feasibility of combining 3 drugs, Revlimid with Doxil and Bevacizumab,and gather preliminary data on the potential activity of the combination in patients with platinum resistant/refractory ovarian cancer.

DETAILED DESCRIPTION:
The combination of Doxil with Avastin has several aspects of interest to ovarian cancer treatment: 1) independent single-agent activity, 2) enhanced localization of Doxil is possible tumoral interstitial pressure via increased half-life (if liposomal egress is diminished) and decreased [42], 3) improved Doxil distribution, and 4) likely favorable toxicity profile since Doxil's only common problematic toxicity is to the skin (palmar-plantar erythrodysesthesia or PPE). Lenalidomide has also antiangiogenic properties, with a different mechanism of action than Avastin. Given the preliminary results of the effect of the combination of Doxil with Avastin, showing an increase in progression-free survival, we are interested in using a new thalidomide analog to maximize the angiogenic inhibition. This study will test the feasibility of combining all 3 drugs, and gather preliminary data on the potential activity of the combination in patients with platinum resistant/refractory ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* EOC patients must be platinum resistant/refractory (see 1.1 for definition) and be considered by the attending physician capable of being treated in this study according to GCP.
* Measurable disease by RECIST criteria or evaluable disease by GCIC criteria
* No prior anthracycline or lenalidomide use, unless the dose received was equal or less than one cycle and the patient did not progress on treatment.
* Subjects must have calculated creatinine clearance > 60ml/min by Cockcroft-Gault formula during the escalation phase.
* Subjects must have calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula during the expansion phase. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance > 30ml/min and < 60ml/min.
* Understand and voluntarily sign an informed consent form.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control.
* No contraindication to anticoagulation

Exclusion Criteria:

* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Concurrent use of other anti-cancer agents or treatments.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* History of thromboembolic event within the last 3 months
* Known hypersensitivity to any component of Avastin

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of the 3 drug combination and recommend a dose for phase II studies. | 6-8 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) after treatment with Revlimid plus Avastin and Doxil. | 6-8 Months
Acute and subacute toxicities of Lenalidomide plus Doxil and Avastin for the treatment of ovarian cancer. | 6-8 Months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Rutledge, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States